CLINICAL TRIAL: NCT03190811
Title: A Prospective Study of Anti-PD-1 Alone or Combined Wih Autologous DC-CIK Cell Therapy in Advanced Solid Tumors
Brief Title: Anti-PD-1 Alone or Combined With Autologous DC-CIK Cell Therapy in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Capital Medical University (Other)
Collaborators: Duke University (Other)
Responsible Party: Principal Investigator, Jun Ren MD, PhD, MD， PhD, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PD1 plus DC-CIK
Record Dates: First submitted 2017-06-15; First posted 2017-06-19 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Neoplasms
Keywords: advanced solid tumor; DC-CIK; anti-PD-1 antibody; immunotherapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anti-PD-1 plus DC-CIK (Experimental)
  Interventions: Biological: Anti-PD-1 plus DC-CIK
- Anti-PD-1 alone (Active Comparator)
  Interventions: Biological: Anti-PD-1 alone

INTERVENTIONS:
Biological: Anti-PD-1 plus DC-CIK — Anti-PD-1 antibody treatment: Patients will receive pembrolizumab 100mg every three weeks until disease progression, unacceptable toxicity or patient refusal.
  DC-CIK Immunotherapy: Mononuclear cells were collected aseptically with blood cell separator composition apheresis, and cultured DC-CIK cells for 10-14 days. Cells were infused back to the patients in 3 times via intravenous infusion .Patients will received at least 2 cycles of DC-CIK Immunotherapy along with 4 dosage of anti-PD-1 antibody treatment. If the evaluation of the treatment is partial response or stable disease, additional cycles were eligible.
  Arms: Anti-PD-1 plus DC-CIK
Biological: Anti-PD-1 alone — Anti-PD-1 antibody treatment: Patients will receive pembrolizumab 100mg every three weeks until disease progression, unacceptable toxicity or patient refusal.
  Arms: Anti-PD-1 alone

SUMMARY:
The purpose of this study is to compare the clinical efficacy and toxicity of anti-PD-1 monoclonal antibody alone with anti-PD-1 monoclonal antibody plus autologous dendritic cells-cytokine induced killer cell (DC-CIK) immunotherapy in advanced tumor patients.Furthermore,to characterize response to therapy we intent to evaluate the role of cell-free DNA (cfDNA) and immune repertoire based on the next generation sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmed advanced or metastatic solid tumors (lung cancer, gastric cancer, renal cancer, bladder cancer, breast cancer, pancreatic cancer, others).
* Patients must have received previously standard therapy for that malignancy or declined to chemotherapy/radiotherapy.
* Estimated life expectancy > 3 months.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0,1 or 2.
* Age 18 to 80.
* Adequate hematologic function, with WBC ≥ 3000/microliter, hemoglobin ≥ 9 g/dL (it is acceptable to have had prior transfusion), platelets ≥ 75,000/microliter; PT-INR <1.5 (unless patient is receiving warfarin in which case PT-INR must be <3), PTT <1.5X ULN
* Adequate renal and hepatic function, with serum creatinine < 1.5 mg/dL, bilirubin < 1.5 mg/dL (except for Gilbert's syndrome which will allow bilirubin ≤ 2.0 mg/dL), ALT and AST ≤ 2.5 x upper limit of normal.

Exclusion Criteria:

* Patients with a history of autoimmune disease, such as but not restricted to, inflammatory bowel disease, systemic lupus erythematosus, ankylosing spondylitis, scleroderma, or multiple sclerosis. Autoimmune related thyroid disease and vitiligo are permitted.
* Patients with serious intercurrent chronic or acute illness, such as cardiac disease (NYHA class III or IV), hepatic disease, or other illness considered by the Principal Investigator as unwarranted high risk for investigational drug treatment.
* Patients with a medical or psychological impediment to probable compliance with the protocol should be excluded.
* Concurrent (or within the last 5 years) second malignancy other than non melanoma skin cancer, cervical carcinoma in situ, controlled superficial bladder cancer, or other carcinoma in situ that has been treated.
* Presence of an active acute or chronic infection including: a urinary tract infection, HIV (as determined by ELISA and confirmed by Western Blot). Patients with HIV are excluded based on immuno-suppression, which may render them unable to respond to the vaccine; patients with chronic hepatitis are excluded because of concern that hepatitis could be exacerbated by the injections.
* Patients on chronic steroid therapy (or other immuno-suppressives, such as azathioprine or cyclosporin A) are excluded on the basis of potential immune suppression. Patients must have had 6 weeks of discontinuation of any steroid therapy (except that used as pre-medication for chemotherapy or contrast-enhanced studies or for acute treatment (<5 days) of intercurrent medical condition such as a gout flare) prior to enrollment.
* Pregnant and nursing women should be excluded from the protocol since this research may have unknown and harmful effects on an unborn child or on young children. If the patient is sexually active, the patient must agree to use a medically acceptable form of birth control while receiving treatment and for a period of 4 months following the last vaccination therapy. It is not known whether the treatment used in this study could affect the sperm and could potentially harm a child that may be fathered while on this study.
* Patients with acute or chronic skin disorders that will interfere with injection into the skin of the extremities or subsequent assessment of potential skin reactions will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2023-06 (Actual)

PRIMARY OUTCOMES:
Overall survival of the participants(OS) | 24 months
  From starting date of anti-PD-1 antibody treatment until date of death from any cause

SECONDARY OUTCOMES:
Progression-free survival of the participants(PFS) | 24 months
  From starting date of anti-PD-1 antibody treatment until date of until the date of first documented disease progression or date of death from any cause, whichever comes first
The changes in immune-response specific patient-reported outcomes(irPRO) | 24 months
  To assess the irPRO scale ratings prior to and after the cancer immunotherapy
Treatment-related adverse events | 24 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
The changes in patient self-reported quality of life | 24 months
  To assess the EORTC QLQ-C30 scale ratings prior to and after the cancer immunotherapy

OTHER OUTCOMES:
Exploratory biomarkers | 24 months
  To investigate the relationship of ctDNA,tumor related antigen peptides, T cell metaboic activity，and microbial bacteria with clincial outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Capital Medical University Cancer Center/Beijing Shijitan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided